CLINICAL TRIAL: NCT06044636
Title: Early Digi-physical Support During Breastfeeding Initiation Linked to Continued Support at the Breastfeeding Clinic
Brief Title: Early Digi-physical Support During Breastfeeding Initiation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marina Taloyan, Associate professor, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BREASTFEEDING
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Breastfeeding; Self Efficacy; Breastfeeding Duration; Depression
Keywords: Breastfeeding; Depression; Primary Healthcare; Digi-physical; Self-Efficacy
MeSH Terms: conditions — Breast Feeding; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digi-physical breastfeeding counceling (Active Comparator): Interventions: Digi-physical breastfeeding counseling
  * At discharge from the maternity ward: contact with lactation consultant (breastfeeding support and care) via the support hotline with chat as soon as questions or problems arise. The hotline will be available during the whole project period.
  * After discharge from the maternity ward: pediatric nurse from Child Health Care Unit (CHC) will contact families and make a home visit (physical or digital), giving extended lactation advice and support. Additional home visits if needed.
  * After discharge until one year after childbirth: the possibility of getting into contact with specialized lactation consultant/nurse at lactation counseling units if needed.
  Intervention type: Chatt via Application Alltid Öppet owned by Region Stockholm.
  The intervention group will follow current healthcare routines in the Region Stockholm and will get access to an evidence-based information package about breastfeeding from pregnancy week 20.
  Interventions: Other: Digi-physical breastfeeding support
- Usual care with physical visits (No Intervention): Title: Usual care with physical visits The control group will follow current healthcare routines in the Region Stockholm and will get access to an evidence-based information package about breastfeeding from pregnancy week 20.

INTERVENTIONS:
Other: Digi-physical breastfeeding support — * Breastfeeding support after birth is provided via chat
  * Extended home visits by a pediatric nurse after discharge from the maternity ward
  * Extra support from a lactation counselor when needed after discharge until one year after childbirth
  Other Names: breastfeeding counceling via chatt function
  Arms: Digi-physical breastfeeding counceling

SUMMARY:
The purpose of this Randomized Controlled Trial is to develop and evaluate a digi-physical intervention within primary health care lactation counselling and breastfeeding support to promote exclusive breastfeeding rates during the first 6 months after birth and to prevent depressive symptoms.

The project addresses parents during pregnancy week 20 and 32 and will continue during the infant's first year of life. All participants will get access to an evidence-based information package (theory and practical advises) during pregnancy.

Study aim is to develop and evaluate digital evidence-based information materials and continuous support for both parents in order to increase prevalence of exclusive breastfeeding and duration as well as decreasing the risks of symptoms of post-partum depression.

DETAILED DESCRIPTION:
The project design is a single-blind randomized controlled trial.

The intervention group will receive:

* Digital support by chat with a lactation consultant for immediate breastfeeding support two-three weeks after delivery
* Extended home visits by pediatric nurses providing extra knowledge and support about lactation
* Extra support by health care providers educated in lactation counseling when needed.

More specific purposes are:

* Compare the prevalence of exclusive breastfeeding until 6 months and duration of breastfeeding up to one year between the intervention and the control group. (Primary outcome)
* Compare prevalence of depression symptoms between the intervention and control group. (Secondary outcome)
* Strengthening parents' self-efficacy in breastfeeding their child.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant or partner of a person who is pregnant in pregnancy week 20-32
* All parents with language skills enabling them to fill out questionnaires, participate in interviews and read information.
* Being resident in Stockholm Region

Exclusion Criteria:

* Parents without adequate Swedish language skills
* Parents resident outside the Stockholm Region

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding at 6 months and duration of breastfeeding | From birth until child is one year old
  Compare the prevalence of exclusive breastfeeding until 6 months and duration of breastfeeding up to one year between the intervention and the control group

SECONDARY OUTCOMES:
Prevalence of depression symptoms | From birth until child is one year old
  Compare prevalence of depression symptoms between intervention and control group 6-8 weeks after births and 6 plus 12 months after birth.

OTHER OUTCOMES:
Parents' self-efficacy breastfeeding their child | From birth until child is one year old
  Compare how parents' self-efficacy breastfeeding their child is improved

CONTACTS AND LOCATIONS:
Overall Officials: Marina Taloyan, Associate Prof., Principal Investigator — Region Stockholm
Locations (1):
- Region Stockholm/Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No